CLINICAL TRIAL: NCT03926715
Title: Prevalence of Malnutrition in Surgery
Acronym: PROMIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Società Italiana di Nutrizione Clinica e Metabolismo (Other)
Collaborators: Campus Bio-Medico University (Other); University of Roma La Sapienza (Other); Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor
Other Study IDs: 01
Record Dates: First submitted 2018-03-17; First posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Malnutrition; Surgery; Cancer
Keywords: Malnutrition; Post-operative complication
MeSH Terms: conditions — Malnutrition; Neoplasms | interventions — Nutritional Status

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nutritional status

SUMMARY:
Nutritional disorders are highly prevalent in gastrointestinal cancer patients undergoing surgery and have shown to contribute significantly in short, mid and long-term clinical outcome. Although increasing evidence and expert suggestions there is still inadequate awareness about the clinical relevance of nutritional and metabolic alterations in surgical oncologic patients.

DETAILED DESCRIPTION:
Nutritional disorders are highly prevalent in cancer patients and have shown to contribute significantly in short-, mid- and long-term clinical outcome. The prevalence of malnutrition is reported between 25% and over 70% based on nutritional assessments. Nutritional disorders represent an important risk factor for the occurence of postoperative complications.

Main obstacles to improving nutritional care include lack of awareness for the problem among the general public and lack of awareness among decision makers and even care providers.

Considering the high prevalence of malnutrition and its repercussions in patient morbidity-mortality and healthcare cost, nutritional screening measures must be included in an integrated nutritional care plan for patients before surgery and while in the hospital.

The PRoMiS study was conceived to quantify nutritional disorders among gastrointestinal cancer patients undergoing surgery in Italy. The data obtained will contribute to increase the awareness of nutritional disorders among oncology surgical patients and their impact on clinical outcome, favoring the inclusion of the initial assessment of nutritional status before surgery and of the nutritional intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are candidates for surgery for gastrointestinal cancer (esophagus, stomach, small intestine, pancreas, biliary tract, colon, rectum, liver)
* Diagnosis of malignant solid tumor
* Age> 18 years
* Informed consent

Exclusion Criteria:

* Uncontrolled metabolic disorders
* Uncompensated heart failure
* Severe psychiatric disorders
* Appropriate logistical support for participation in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are candidates for surgery for gastrointestinal cancer (esophagus, stomach, small intestine, pancreas, biliary tract, colon, rectum, liver)
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2017-01-06 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Malnutrition | Pre-operative
  Malnutrition will be assessed by Malnutrition Universal Screening Tool (MUST)

SECONDARY OUTCOMES:
Post-operative complications | Hospital discharge (10-15 days)
  Incidence of pneumonia, sepsis and dehiscence of the surgical wound.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Coppola, Principal Investigator — Campus Bio-Medico of Rome
Locations (8):
- Italy (8):
  - Pof. Romario Fumagalli, Brescia
  - Leonardo De Meo, Catania
  - Claudio Pedrazzi, Reggio Emilia
  - Roberto Coppola, Rome
  - Antonio Gasbarrini, Rome
  - Roberto Caronna, Rome
  - Amilcare Parisi, Terni
  - Giovanni de Manzoni, Verona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Garcia GH, Fu MC, Dines DM, Craig EV, Gulotta LV. Malnutrition: a marker for increased complications, mortality, and length of stay after total shoulder arthroplasty. J Shoulder Elbow Surg. 2016 Feb;25(2):193-200. doi: 10.1016/j.jse.2015.07.034. Epub 2015 Oct 9. PMID 26456427
- [Result] Culebras JM. Malnutrition in the twenty-first century: an epidemic affecting surgical outcome. Surg Infect (Larchmt). 2013 Jun;14(3):237-43. doi: 10.1089/sur.2013.9993. Epub 2013 May 15. No abstract available. PMID 23676121
- [Result] Mahdi H, Jernigan AM, Aljebori Q, Lockhart D, Moslemi-Kebria M. The impact of obesity on the 30-day morbidity and mortality after surgery for endometrial cancer. J Minim Invasive Gynecol. 2015 Jan;22(1):94-102. doi: 10.1016/j.jmig.2014.07.014. Epub 2014 Jul 24. PMID 25064420
- [Result] Hebuterne X, Lemarie E, Michallet M, de Montreuil CB, Schneider SM, Goldwasser F. Prevalence of malnutrition and current use of nutrition support in patients with cancer. JPEN J Parenter Enteral Nutr. 2014 Feb;38(2):196-204. doi: 10.1177/0148607113502674. PMID 24748626
- [Result] Ejaz A, Spolverato G, Kim Y, Poultsides GA, Fields RC, Bloomston M, Cho CS, Votanopoulos K, Maithel SK, Pawlik TM. Impact of body mass index on perioperative outcomes and survival after resection for gastric cancer. J Surg Res. 2015 May 1;195(1):74-82. doi: 10.1016/j.jss.2014.12.048. Epub 2014 Dec 31. PMID 25619462
- [Result] Muscaritoli M, Molfino A, Gioia G, Laviano A, Rossi Fanelli F. The "parallel pathway": a novel nutritional and metabolic approach to cancer patients. Intern Emerg Med. 2011 Apr;6(2):105-12. doi: 10.1007/s11739-010-0426-1. Epub 2010 Jul 2. PMID 20596799
- [Result] Cederholm T, Bosaeus I, Barazzoni R, Bauer J, Van Gossum A, Klek S, Muscaritoli M, Nyulasi I, Ockenga J, Schneider SM, de van der Schueren MA, Singer P. Diagnostic criteria for malnutrition - An ESPEN Consensus Statement. Clin Nutr. 2015 Jun;34(3):335-40. doi: 10.1016/j.clnu.2015.03.001. Epub 2015 Mar 9. PMID 25799486
- [Result] Fearon K, Strasser F, Anker SD, Bosaeus I, Bruera E, Fainsinger RL, Jatoi A, Loprinzi C, MacDonald N, Mantovani G, Davis M, Muscaritoli M, Ottery F, Radbruch L, Ravasco P, Walsh D, Wilcock A, Kaasa S, Baracos VE. Definition and classification of cancer cachexia: an international consensus. Lancet Oncol. 2011 May;12(5):489-95. doi: 10.1016/S1470-2045(10)70218-7. Epub 2011 Feb 4. PMID 21296615
- [Result] Muscaritoli M, Anker SD, Argiles J, Aversa Z, Bauer JM, Biolo G, Boirie Y, Bosaeus I, Cederholm T, Costelli P, Fearon KC, Laviano A, Maggio M, Rossi Fanelli F, Schneider SM, Schols A, Sieber CC. Consensus definition of sarcopenia, cachexia and pre-cachexia: joint document elaborated by Special Interest Groups (SIG) "cachexia-anorexia in chronic wasting diseases" and "nutrition in geriatrics". Clin Nutr. 2010 Apr;29(2):154-9. doi: 10.1016/j.clnu.2009.12.004. Epub 2010 Jan 8. PMID 20060626